CLINICAL TRIAL: NCT03294278
Title: Epicardial Ablation in Brugada Syndrome in the Prevention of Sudden Cardiac Death. A Randomized Prospective Follow-up Study.
Brief Title: Epicardial Ablation in Brugada Syndrome to Prevent Sudden Death
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Carlo Pappone, Chief of Arrhythmology Department, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRCCSDonato Brugada-randomized
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Ventricular Arrhythmias and Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation plus ICD (Active Comparator): Epicardial ablation by radio-frequency
  Interventions: Other: ablation plus ICD
- ICD alone (Active Comparator): Implantation of ICD
  Interventions: Other: ablation plus ICD

INTERVENTIONS:
Other: ablation plus ICD — Defibrillator, radio-frequency catheter ablation

SUMMARY:
A total of 150 patients will be randomized to perform catheter ablation or not in a 2:1 fashion in selected patients with Brugada-related symptoms (Ablation+ICD arm 105 patients vs ICD only 45 patients).

DETAILED DESCRIPTION:
The main purpose of this trial is to develop evidence-based curative treatment with optimal net benefit for patients with Brugada syndrome. As recent non-randomized pilot studies and scarce case reports documented the potential benefit of epicardial ablation, patients in this trial will be randomized to epicardial catheter ablation of the regions exhibiting abnormally prolonged and fragmented electrograms in the right ventricular outflow tract plus continued implanted cardioverter defibrillator therapy (ablation arm) or continued implanted cardioverter defibrillator therapy (control arm).

Survival from any ventricular arrhythmia (VA) recurrence will be considered as primary endpoint.

A projected 150 patients will be enrolled and randomized to receive ablation or not in a 2:1 fashion (Ablation+ICD arm 105 patients vs ICD only 45 patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by Brugada Syndrome diagnosed according to 2013 HRS/EHRA/APHRS
* Consensus document criteria
* The patient received at least 1 appropriate ICD shock.
* Documentation of any previous ventricular arrhythmia (VA) in the form of VT, non-sustained VT, non-sustained VF, RVOT PVC with a daily burden >10000;
* Age ≥ 18;
* Willingness to attend follow-up examinations;
* Written informed consent for participation in the trial.

Exclusion Criteria:

* A patient who does not meet inclusion criteria;
* Pregnancy or breast-feeding (which would exclude an ablation procedure);
* Contraindications to general anesthesia or epicardial ablation;
* Life expectancy < 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-09-10 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival from any VA recurrence will be considered as primary endpoint | 2 years after ablation
  NO ventricular arrhythmia recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, Principal Investigator — IRCCS Policlinico San Donato Milan, Italy
Locations (1):
- IRCCS Policlinico S. Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pappone C, Ciconte G, Vicedomini G, Micaglio E, Boccellino A, Negro G, Giannelli L, Rondine R, Creo P, Tarantino A, Ballarotto M, Maiolo V, Ciaccio C, Manuello R, Locati ET, Mazza BC, Vecchi M, Calovic Z, Anastasia L. Epicardial ablation in high-risk Brugada syndrome to prevent ventricular fibrillation: results from a randomized clinical trial. Europace. 2025 May 7;27(5):euaf097. doi: 10.1093/europace/euaf097. PMID 40401314